CLINICAL TRIAL: NCT04192903
Title: Chidamide Combined With Cisplatin for Relapsed or Metastatic Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1910208-9
Record Dates: First submitted 2019-12-07; First posted 2019-12-10 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide combined with Cisplatin (Experimental): Chidamide: 30mg,PO,biw one week before cycle 1 treatment
  Combined treatment period:
  Cisplatin 75mg/m2 ivgtt D1 Chidamide :20mg PO Biw, 2 week on , 1 week off Patients whose efficacy was evaluated as Complete Response (CR) / Partial Response (PR) / Stable Disease (SD) after the end of the combined treatment period received maintenance treatment with chidamide combined with cisplatin reduction.
  Maintenance treatment period:
  Cisplatin 25mg/m2 ivgtt D1 Chidamide :20mg PO Biw, 2 week on , 1 week off
  Interventions: Drug: Chidamide combined with Cisplatin

INTERVENTIONS:
Drug: Chidamide combined with Cisplatin — Chidamide: 30mg,PO,biw one week before cycle 1 treatment Cisplatin 75mg/m2 ivgtt D1 Chidamide :20mg PO Biw, 2 week on , 1 week off

SUMMARY:
The goal of this clinical trial is to evaluate therapeutic efficacy and safety of Chidamide combined with Cisplatin for relapsed or metastatic triple-negative breast cancer.

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC), the most difficult-to-treat breast cancer subtype, lacks well-defined treatment options. This is a prospective, single-center, one-arm, open-label, phase II clinical trial evaluating the efficacy and safety of chidamide in combination with cisplatin in subjects with relapsed or metastatic triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 years (including cutoff value).
2. Patients with recurrent or metastatic breast cancer , histologically proven invasive breast carcinoma with triple negative receptor status (Estrogen receptor, Progesterone receptor and HER2 negative by IHC and FISH) by histopathology in Department of Pathology, Fudan University Cancer Center, Local recurrence needs to be confirmed by the physician that is unresectable.
3. Prior treatment:Previously received no more than 1prior lines of systemic chemotherapy for metastatic breast cancer, and progressed after treatment, chemotherapy regimen did not contain cisplatin or did not demonstrate cisplatin resistance (disease progression during the cisplatin treatment period or within 3 months after completion);
4. At least one extracranial measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
5. Eastern Cooperative Oncology Group Performance Status of 0-1.
6. Life expectancy ≥ 3 months.
7. Adequate function of major organs meets the following requirements (no blood components and cell growth factors have been used within 14 days before randomization):

   Neutrophils ≥ 1.5×10^9/L Platelets ≥ 90×10^9/L Hemoglobin ≥ 90g/L Total bilirubin≤ 1.5 × the upper limit of normal (ULN) ALT and AST ≤ 2.5 × ULN BUN and Cr ≤ 1.5 × ULN Left ventricular ejection fraction (LVEF) ≥ 50% QTcF(Fridericia correction) ≤ 470 ms International normalized ratio(INR)≤1.5 × ULN，activated partial thromboplastin time(APTT) ≤ 1.5 × ULN
8. Subjects voluntarily joined the study, signed informed consent.

Exclusion Criteria:

1. Previously received any HDAC inhibitor treatment.
2. The subject has untreated central nervous system (CNS) metastases.
3. Patients who have undergone systemic, radical brain or meningeal metastasis (radiotherapy or surgery), but have been confirmed to have been stable for at least 4 weeks, and who have stopped systemic hormonal therapy for more than 2 weeks without clinical symptoms can be included.
4. Previously received more than 2 lines of systemic chemotherapy for metastatic breast cancer.
5. There are ascites, pleural effusion, pericardial effusion with clinical symptoms at baseline, those who need drainage, or those who have undergone drainage of serous effusion within 4 weeks before the first dose.
6. Inability to swallow, intestinal obstruction or other factors affecting the administration and absorption of the drug.
7. Received systemic therapy such as chemotherapy, molecular targeted therapy or other clinical trial drugs within 4 weeks before enrollment;
8. Patients with other malignant tumors within 5 years or at the same time( except for cured skin basal cell carcinoma and cervical carcinoma in situ).
9. Have undergone major surgical procedures or significant trauma within 4 weeks prior to randomization, or are expected to undergo major surgery.
10. Have a history of allergies to the drug components of this regimen.
11. Patients with active HBV and HCV infection; stable hepatitis B after drug treatment (HBV virus copy number is higher than the upper limit of reference value) and cured hepatitis C patients (HCV virus copy number exceeds the lower limit of detection method) can be included.
12. History of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disease, history of organ transplantation.
13. History of cardiac dysfunction, include(1)angina (2)clinical significant arrythmia or require drug intervention (3)myocardial infarction (4)heart failure (5) other cardiac dysfunction (judged by the physician); any cardiac or nephric abnormal ≥ grade 2 found in screening.
14. Female patients who are pregnancy, lactation or women who are of childbearing potential tested positive in baseline pregnancy test. Childbearing female who refuse to accept any contraception practice during the treatment period and for at least 8 weeks after the last dose of chemotherapy.
15. Determined by the physician, any serious coexisting disease might be harmful to the patient's safety or avoid the patients from accomplishing the treatment(e.g serious hypertension, diabetes, thyroid dysfunction, active infection etc.).
16. History of neurological or psychiatric disorders, including epilepsy or dementia.
17. The investigator determined who was not suitable for the study.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2019-12-25 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | From the day of treatment to the date of first documented progression，up to 18 months after the last patient's enrollment
  Defined as numbers of patients achieved complete response and partial response of treatment

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From the day of treatment to the date of first documented progression，up to 18 months after the last patient's enrollment
  Defined as the time from randomization until objective tumor progression or death
Overall survival (OS) | From the day of treatment to the date of first documented progression，up to 18 months after the last patient's enrollment
  Defined as from the date of inclusion to date of death, irrespective of cause
Duration of remission (DOR) | From the day of treatment to the date of first documented progression，up to 18 months after the last patient's enrollment
  Defined as from date of complete remission to date of progression, relapse, or death from any cause
Clinical Benefit Rate (CBR) | From the day of treatment to the date of first documented progression，up to 18 months after the last patient's enrollment
  Proportion of participants with a clinical benefit (CB), defined as an objective response (CR or PR), or stable disease for at least 24 weeks, as determined by the Investigator through the use of RECIST v1.1.
Adverse event(AE) | From the day of treatment to the date of first documented progression，up to 18 months after the last patient's enrollment
  Adverse event related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: xichun Hu,MD, Study Director — Fudan University; Jian Zhang,MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China